CLINICAL TRIAL: NCT03719417
Title: A Biologic Joint Replacement Strategy to Treat Patients With Severe Knee Trauma and Post-Traumatic Osteoarthritis (Expansion)
Brief Title: A Biologic Joint Replacement Strategy for Knee Trauma and Post-Traumatic Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, James Stannard, Professor, Orthopedic Surgery, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011153
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Knee Osteoarthritis; Post-traumatic Osteoarthritis
Keywords: Knee Pain
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unicompartmental Biologic Arthroplasty (Active Comparator): Subject will be receiving a unicompartmental biologic arthroplasty only
  Interventions: Procedure: Unicompartmental Biologic Arthroplasty
- Extensive Biologic Arthroplasty (Active Comparator): Subject will be receiving a unicompartmental biologic arthroplasty with at least one additional surface in another compartment being replaced concurrently.
  Interventions: Procedure: Extensive Biologic Arthroplasty

INTERVENTIONS:
Procedure: Unicompartmental Biologic Arthroplasty — Unicompartmental Biologic Arthroplasty surgery.
  Arms: Unicompartmental Biologic Arthroplasty
Procedure: Extensive Biologic Arthroplasty — Unicompartmental Biologic Arthroplasty surgery with an additional surface being replaced concurrently
  Arms: Extensive Biologic Arthroplasty

SUMMARY:
Participants will be enrolled in a prospective clinical trial to assess outcomes in 2 cohorts of patients undergoing unicompartmental versus more extensive biologic OCA transplantation of the knee using MOPSTM-preserved allografts (including menisci), anatomically-shaped allografts, autogenous bone marrow aspirate concentrate (BMC)-treated donor bone, and treatment-specific postoperative rehabilitation.

DETAILED DESCRIPTION:
With IRB approval, patients will be enrolled in a prospective clinical trial to assess outcomes in 2 cohorts of patients undergoing unicompartmental versus more extensive biologic OCA transplantation of the knee using MOPSTM-preserved allografts (including menisci), anatomically-shaped allografts, autogenous bone marrow aspirate concentrate (BMC)-treated donor bone, and treatment-specific postoperative rehabilitation. Demographic and operative data will be collected. Outcome assessments will include VAS pain, IKDC, SANE, Tegner and PROMIS Mobility for knee at 6 months and yearly after surgery. In addition, serial limb alignment measurements, ultrasonographic assessments of meniscal location and integrity, quantitative MRIs for cartilage composition, and serum and urine biomarkers for treatment monitoring will be performed. All complications and re-operations will be recorded. OCA survival will be determined based on maintenance of acceptable levels of pain and function and/or need for revision surgery or total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Grade IV changes in the articular cartilage of the femoral condyle and tibial plateau and meniscal pathology in the medial or lateral femorotibial joint (unicompartmental) or unicompartmental and other femoral condyle, tibial plateau, trochlea and/or patella.
* Between the age of 18-55

Exclusion Criteria:

* Acute injury to any other part of the affected lower extremity
* Inability to comply with protocol
* BMI greater than 40
* The subject is either pregnant or a prisoner
* Currently involved in worker's compensation case at the time of enrollment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
VAS Pain Score (Visual Analog Scale) | 12 Months
  This pain score is between 0 and 10, with 0 being no pain and 10 being the worst pain

SECONDARY OUTCOMES:
International Knee Documentation Committee Score (IKDC) | 12 Months
  This score looks at pain and function scores. 0 is the lowest score and 100 is the highest function score.
Single Assessment Numeric Evaluation (SANE) score | 12 Months
  This score looks at what the patient rates their knee with 100% being normal, and 0% being as far from normal as possible
PROMIS Mobility | 12 Months
  This looks at mobility and function on a scale of 14.1 to 61.7 with higher scores equaling higher mobility

CONTACTS AND LOCATIONS:
Overall Officials: James Stannard, MD, Principal Investigator — University of Missouri, Department of Orthopaedic Surgery
Locations (1):
- Missouri Orthopaedic Institute, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No